CLINICAL TRIAL: NCT04059757
Title: Fecal Microbiota Transplantation For The Treatment Of Gastro-Intestinal Acute Graft Versus Host Disease
Brief Title: Fecal Microbiota Transplantation For The Treatment Of Gastro-Intestinal Acute GVHD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Drugs unavailable
Sponsor: Leland Metheny (Other)
Responsible Party: Sponsor-Investigator, Leland Metheny, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE4Z19
Record Dates: First submitted 2019-08-07; First posted 2019-08-16 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Gastro-Intestinal Acute Graft Versus Host Disease (GI-aGVHD)
Keywords: Graft Versus Host Disease (GVHD)
MeSH Terms: conditions — Graft vs Host Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: The study follows R. Simon's minimax two-stage phase II design with type I error of 0.05 and power of 80%. Ten participants will be enrolled on stage one. If there are 2 or less responses, the trial will be stopped and the treatment will be considered less than 60% effective for this patient population. If there are 3 or more responses, 7 additional patients will be enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fecal Microbiota Transplantation (FMT) (Experimental): One dose of FMT equal to 30 capsules will be administered on day 1 of a 28 day cycle. Steroids and routine GVHD prophylaxis medications and antibiotics may be administered concurrently with FMT therapy.
  Participants will be followed for 28 days following completion of the FMT dose or protocol defined outcome.
  aGVHD will be treated as per standard of care.
  Interventions: Biological: Fecal Microbiota Transplantation (FMT)

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation (FMT) — 1 dose = 30 capsules on day 1 of Fecal Microbiota Transplantation

SUMMARY:
Gastro-Intestinal Acute Graft Versus Host Disease (GI-aGVHD) is a complication of allogeneic stem cell transplant which is usually treated with steroids. You are being asked to take part in this study because you have recently been diagnosed with GI-GVHD. The standard of care for GI-aGVHD is steroids. When aGVHD does not respond to steroids it is described as steroid-refractory aGVHD. There is no standard therapy for steroid-refractory GI-aGVHD.

This study is a Phase II study. The main goal of a Phase II study is to see the efficacy and what side effects are seen with FMT as a treatment for GVHD.

Fecal Microbiota Transplantation (FMT) is the transfer of fecal material from a healthy donor to a patient in order to restore the diversity of the intestinal microbiota. FMT is currently indicated for the treatment of recurrent Clostridium Difficile infection.

FMT is considered experimental in this study, meaning it is not approved by the FDA for the treatment of GVHD.

ELIGIBILITY:
Inclusion Criteria:

* One of the following diagnosis:
* High risk aGVHD (either biopsy proven or clinical diagnosed) (see Appendix B & C) as defined by either:

  * Lower gastrointestinal (GI) stage 3+
  * Hyper-acute GVHD as defined by aGVHD of the GI tract within the first 14 days of transplant AND
  * Subjects with treatment-naive acute GVHD as defined as those who have not received previous systemic treatment for acute GVHD, except for a maximum of 7 days of no less than 1 mg/kg/day of methyl-prednisolone (or equivalent dose of prednisone).

OR:

* Steroid refractory aGVHD of the GI tract (either biopsy proven or clinical diagnosed) as defined by:

  * no response to steroid treatment (minimum daily dose: 2 mg/kg methyl-prednisolone or equivalent) lasting at least 7 days, or
  * progression of at least one grade within the first 72 h of treatment
* ECOG Performance status < 3
* Patients who underwent an allogeneic hematopoietic stem cell transplantation from any donor source.
* Patients who are able stop prophylactic antibiotics during the treatment period
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Active malignancy
* Patients with any concurrent uncontrolled clinically significant medical condition including active infection, laboratory abnormality, or psychiatric illness which could place the patient at unacceptable risk of study treatment.
* Pregnant or breastfeeding women
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the subject; or interfere with interpretation of study data.
* Known allergies, hypersensitivity, or intolerance to any of the study medications, excipients, or similar compounds
* Patients with any severe gastrointestinal condition other than GI-GVHD.
* Inability (e.g. dysphagia) to or unwilling to swallow capsules
* Active gastrointestinal infection at time of enrollment
* Known or suspected toxic megacolon and/or known small bowel ileus
* Major gastrointestinal surgery (e.g. significant bowel resection) within 3 months before enrollment. This does not include appendectomy or cholecystectomy
* History of total colectomy or bariatric surgery
* Concurrent intensive induction chemotherapy, radiation therapy or biological treatment for active malignancy
* Unable or unwilling to comply with protocol requirements
* Expected life expectancy < 6 months
* Patients who have CMV >2,000 copies/mL of whole blood or EBV >2,000 copies/mL of whole blood.

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing toxicity | up to 6 months from start of treatment
  Toxicity is defined as:
  * Any bacterial or fungal infection that can be definitely attributed to FMT.
  * Any grade 3 or more adverse event that occurs during or immediately after receiving the treatment and is definitely attributed to FMT.
Efficacy of FMT therapy in high risk and in steroid refractory GI-aGVHD as defined as number of responses at day 28 (+/- 3 days) post FMT treatment | 28 days (+/- 3 days) post FMT treatment
  Response will be determined from the maximum GI-aGVHD stage and grade at day 28 (+/- 3 days) post FMT treatment. Response will be determined by P.I and a second physician.
  * Complete response (CR) is defined as the complete resolution of GI aGVHD symptoms, without secondary GVHD therapy.
  * Partial response (PR) is defined as improvement without complete resolution and without worsening of GI aGVHD, without secondary aGVHD therapy.
  * No response (NR) is defined as the same grade of GVHD, progression, death, or the addition of secondary GVHD therapy.
  * Progression is defined as worsening GI aGVHD.

SECONDARY OUTCOMES:
Non-relapse mortality (NRM) as measured by percentage of participants who die not related to relapse | up to 6 months from start of treatment
  Non-relapse mortality (NRM) as measured by percentage of participants who die not related to relapse
Relapse as measured by percentage of participants who relapse | up to 6 months from start of treatment
  Relapse as measured by percentage of participants who relapse
Relapse-related mortality as measured by percentage of participants with death related to relapse | up to 6 months from start of treatment
  Relapse-related mortality as measured by percentage of participants with death related to relapse.
Percentage of participants who develop cGVHD by the end of trial | up to 6 months from start of treatment
  Percentage of participants who develop cGVHD by the end of trial
Overall survival (OS) as measured by percentage of participants who are alive at end of trial | up to 6 months from start of treatment
  Overall survival (OS) as measured by percentage of participants who are alive at end of trial
Percentage of patients who discontinue steroids at the end of the study | up to 6 months from start of treatment
  Percentage of patients who discontinue steroids at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Leland Metheny, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline or influence the results observed from the study.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Investigators who provide a methodologically sound proposal for use of requested data.